CLINICAL TRIAL: NCT02953548
Title: A Randomized, Double-blind, Placebo-controlled Trial to Investigate the Efficacy and Safety of Cannabidiol (CBD; GWP42003-P) in Infants With Infantile Spasms Following an Initial Open-label Pilot Study
Brief Title: Trial of Cannabidiol (CBD; GWP42003-P) for Infantile Spasms (GWPCARE7)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWEP15100 Pilot Phase; 2015-004904-50 (EudraCT Number)
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Results first posted 2020-07-23 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Infantile Spasms
Keywords: GWP42003-P; Cannabidiol
MeSH Terms: conditions — Spasms, Infantile | interventions — Cannabidiol

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GWP42003-P (Experimental): Administered orally, titrating to a target dose of 40 mg/kg/day. Participants continue at the target dose, or the highest tolerated dose up to the target dose, for the remainder of the 2-week treatment period.
  Interventions: Drug: GWP42003-P

INTERVENTIONS:
Drug: GWP42003-P — Clear, colorless to yellow solution containing cannabidiol dissolved in the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring.
  Other Names: CBD; Cannabidiol

SUMMARY:
This trial consists of 3 parts: a pilot safety phase, a pivotal randomized controlled phase, and an open-label extension phase. The pilot phase only will be described in this record. 2 cohorts of 5 participants will be enrolled sequentially. All participants will receive GWP42003-P.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant is aged 6- 24 months (inclusive) in the first cohort or aged 1-24 months (inclusive) in the second cohort, at the time of consent.
* Participant is diagnosed with IS and has failed to respond adequately following treatment with 1 or more approved IS therapies.
* To be considered hypsarrhythmia, as defined for use in the study, the electroencephalography (EEG) background must be slowed and have multifocal spikes. In addition, it must be either high voltage (above 300 µV) or have electrodecrement/discontinuity.

Key Exclusion Criteria:

* Participant is currently taking or has taken clobazam or any mammalian target of rapamycin (mTOR) inhibitor within the 2 weeks prior to the screening visit.
* Participant has a QT interval, corrected for heart rate with Bazett's formula (QTcB), of 460 msec or greater on ECG.
* Participant's caregiver is currently giving or has given recreational or medicinal cannabis, or synthetic cannabinoid-based medications, within the 1 month prior to the screening visit.
* Participant's caregiver is unwilling to abstain from giving the participant (including the participant's mother abstaining themselves, if breastfeeding)recreational or medicinal cannabis, or synthetic cannabinoid-based medications (other than the study drug) during the trial.
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the study drug, such as sesame oil.
* Participant has significantly impaired hepatic function at the screening visit.
* Participant has received an investigational medicinal product as part of a clinical trial within a minimum of 5 half-lives prior to the screening visit.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - The Childrens Hospital of San Antonio, San Antonio, Texas
  - Valley Health Clinical Research, Winchester, Virginia
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Medyczne POMOC, Lodz

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened to assess their eligibility to enter the trial within 7 days prior to the first dose administration.
Groups:
- Cohort 1: GWP42003-P OS: Participants 6 months to 24 months of age received GWP42003-P oral solution (OS) for 14 days. Starting on Day 1 and over the course of 4 days, participants titrated up to a tolerable dose, not to exceed the target dose of 40 milligrams per kilograms per day (mg/kg/day) of GWP42003-P.
- Cohort 2: GWP42003-P OS: Participants 1 month to 24 months of age received GWP42003-P OS for 14 days. Starting on Day 1 and over the course of 4 days, participants titrated up to a tolerable dose, not to exceed the target dose of 40 mg/kg/day of GWP42003-P.
Period: Overall Study
Arm/Group | Cohort 1: GWP42003-P OS | Cohort 2: GWP42003-P OS
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- GWP42003-P OS: Participants received GWP42003-P oral solution (OS) for 14 days. Starting on Day 1 and over the course of 4 days, participants titrated up to a tolerable dose, not to exceed the target dose of 40 mg/kg/day of GWP42003-P.
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (5.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs are defined as all adverse events not present prior to the first investigational medicinal product (IMP) or placebo administration or any event already present that worsened in severity or frequency following IMP.
Time Frame: From signing of informed consent up to Day 15
Population: Safety Analysis Set: all participants who received at least 1 dose of GWP42003-P
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 6

2. Primary Outcome: Number of Participants With Any Low or High Hematology Laboratory Parameter Value
Time Frame: Day 4 and Day 15
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- GWP42003-P OS: Participants received GWP42003-P OS for 14 days. Starting on Day 1 and over the course of 4 days, participants titrated up to a tolerable dose, not to exceed the target dose of 40 mg/kg/day of GWP42003-P.
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 4, Low | 4
  Day 4, High | 4
  Day 15, Low: number analyzed (Participants) | 8
  Day 15, Low | 1
  Day 15, High: number analyzed (Participants) | 8
  Day 15, High | 3

3. Primary Outcome: Number of Participants With Any Low or High Biochemistry Laboratory Parameter Value
Time Frame: Day 4 and Day 15
Population: Safety Analysis Set. Only participants with evaluable data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 4, Low | 7
  Day 4, High | 5
  Day 15, Low: number analyzed (Participants) | 8
  Day 15, Low | 5
  Day 15, High: number analyzed (Participants) | 8
  Day 15, High | 7

4. Primary Outcome: Number of Participant With Any Clinically Relevant Urinalysis Parameter Value
Description: Clinical relevance was determined by the investigator.
Time Frame: Day 4 and Day 15
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 4 | 0
  Day 15 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram Findings
Description: Clinical significance was determined by the investigator.
Time Frame: From signing of informed consent up to Day 15
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 0

6. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: Clinical significance was determined by the investigator.
Time Frame: From signing of informed consent up to Day 15
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 0

7. Primary Outcome: Number of Participants With Clinically Significant Vital Sign Findings
Description: Clinical significance was determined by the investigator.
Time Frame: From signing of informed consent up to Day 15
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 0

8. Secondary Outcome: Number of Participants Free of Clinical Spasms
Description: Clinical spasms were determined by video-electroencephalography (VEEG) for at least 8 hours and up to 24 hours.
Time Frame: Day 15
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 0

9. Secondary Outcome: Percentage of Participants Free of Clinical Spasms
Description: Clinical spasms were determined by VEEG for at least 8 hours and up to 24 hours.
Time Frame: Day 15
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
percentage of participants | 0

10. Secondary Outcome: Number of Participants With Resolution of Hypsarrhythmia
Description: Resolution of hypsarrhythmia was determined by VEEG for at least 8 hours and up to 24 hours.
Time Frame: Day 15
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants | 0

11. Secondary Outcome: Percentage of Participants With Resolution of Hypsarrhythmia
Description: Resolution of hypsarrhythmia was determined by VEEG for at least 8 hours and up to 24 hours.
Time Frame: Day 15
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
percentage of participants | 0

12. Secondary Outcome: Number of Participants Experiencing Spasms and Seizures by Subtype
Description: Caregivers recorded the participant's spasms and seizures by category in a daily diary. Subtypes of spasms and seizures included: clonic, tonic-clonic, myoclonic, focal, and absence.
Time Frame: Day 4 and Day 15
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
Participants
  Day 4, Clonic | 0
  Day 4, Tonic-Clonic | 1
  Day 4, Atonic | 0
  Day 4, Myoclonic | 0
  Day 4, Focal | 1
  Day 4, Absence | 0
  Day 4, Not Done | 0
  Day 15, Clonic | 0
  Day 15, Tonic-Clonic | 0
  Day 15, Atonic | 0
  Day 15, Myoclonic | 0
  Day 15, Focal | 2
  Day 15, Absence | 0
  Day 15, Not Done | 0

13. Secondary Outcome: Average Time to Cessation of Spasms
Description: Analysis could not be conducted for this outcome measure because the study met No Go Criteria. The Pilot Phase concluded after 9 participants completed treatment and demonstrated continued hypsarrhythmia and spasms on follow-up VEEG. The Pivotal Phase was not initiated; however, participants completing the Pilot Phase could roll into the Open Label Extension Phase (NCT02954887) for up to 1 year.
Time Frame: Day 1 to start of Open-label Extension (OLE) Phase
Population: Safety Analysis Set
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 0

14. Secondary Outcome: Caregiver Clinical Global Impression of Change (CGIC)
Description: The CGIC is a single-question assessment completed by the caregiver. The question assessed the status of the participant's condition since treatment start. The caregiver provided a rating on a 7-point scale from 1 (very much improved) to 7 (very much worse).
Time Frame: Day 15
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
participants
  Very Much Improved | 1
  Much Improved | 0
  Slightly Improved | 7
  No Change | 1
  Slightly Worse | 0
  Much Worse | 0
  Very Much Worse | 0
  Not Done | 0

15. Secondary Outcome: Physician Global Impression of Change (PGIC)
Description: The PGIC is a single-question assessment completed by the investigator. The question assesses the status of the participant's condition since treatment start. The investigator provided a rating on a 7-point scale from 1 (very much improved) to 7 (very much worse).
Time Frame: Day 15
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | GWP42003-P OS
Number analyzed (Participants) | 9
participants
  Very Much Improved | 0
  Much Improved | 1
  Slightly Improved | 5
  No Change | 3
  Slightly Worse | 0
  Much Worse | 0
  Very Much Worse | 0
  Not Done | 0

16. Secondary Outcome: Number of Responders
Description: A responder is defined as a participant experiencing a resolution of hypsarrhythmia and free of spasms. Testing for responders was conducted by VEEG for at least 8 hours and up to 24 hours.
Time Frame: Baseline to Day 15
Population: Safety Analysis Set
Measure: Number; unit: responders
Arm/Group | Cohort 1: GWP42003-P OS | Cohort 2: GWP42003-P OS
Number analyzed (Participants) | 5 | 4
responders | 0 | 0

17. Secondary Outcome: Percentage of Responders
Description: as for outcome 16
Time Frame: Baseline to Day 15
Population: Safety Analysis Set
Measure: Number; unit: responders
Arm/Group | Cohort 1: GWP42003-P OS | Cohort 2: GWP42003-P OS
Number analyzed (Participants) | 5 | 4
responders | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to Day 15
Description: Treatment-emergent adverse events (TEAEs) were collected in members of the Safety Population, comprised of all participants who received at least 1 dose of GWP42003-P. TEAEs are defined as all adverse events not present prior to the first investigational medicinal product (IMP) or placebo administration or any event already present that worsened in severity or frequency following IMP.
Arm/Group | GWP42003-P OS
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P OS (N=9)
Status epilepticus (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P OS (N=9)
Application site erosion (General disorders) | 1
Irritability (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Somnolence (Nervous system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 2

LIMITATIONS AND CAVEATS:
This study met No Go Criteria. The Pilot Phase concluded after 9 participants completed treatment, and the Pivotal Phase was not initiated. Participants completing the Pilot Phase could roll into the Open Label Extension Phase for up to 1 year.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-09-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT02953548/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT02953548/SAP_001.pdf